CLINICAL TRIAL: NCT02322125
Title: Restoring Walking With a Powered Exoskeleton After Complete and Sever Incomplete Spinal Cord Injury
Brief Title: Restoring Walking With a Powered Exoskeleton After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00036789
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Spinal Cord Injury
Keywords: walking; locomotion; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ReWalk training (Experimental): ReWalk exoskeleton training: 1.5 hr/day, 4 days/week, for 12-14 weeks (approximately 50 training sessions). Participants will progress through the following: sit-to-stand, stand-to-sit, standing balance and weight shift, walking on smooth ground, stopping, turning while walking, walking on rough ground, ascending and descending slopes, ascending and descending steps and curbs.
  Interventions: Device: ReWalk

INTERVENTIONS:
Device: ReWalk — Intensive training with the ReWalk to negotiate smooth ground, rough terrain indoors and outdoors, ascending and descending slopes and steps, in a home setting and in the community.

SUMMARY:
Powered exoskeletons have emerged recently, promising to offer walking to individuals with severe spinal cord injury who are unable to walk. We will use the ReWalk exoskeleton to train walking in individuals with chronic, severe spinal cord injury (SCI). We will determine the characteristics of individuals who most benefit from such training, and identify the neuroplasticity induced by the training. We will further determine the feasibility of the ReWalk for home and community ambulation.

DETAILED DESCRIPTION:
A prospective, pilot, cohort study design will recruit participants to train intensively for a 3 month period. The training sessions will be documented in detail, including number of steps taken, speed of walking, distance of walking. Once walking speed has plateaued, we will evaluate the feasibility of using the device in a home-like environment and in the community.

At the end of this study, we will have a good idea of the capability of the ReWalk to assist walking in those with severe spinal cord injury. We will better understand which individuals are most likely to benefit from the ReWalk. We will know how training in the ReWalk changes the neural connections between the brain and the spinal cord so that we can better guide the training protocol. Finally, we will identify limitations of the ReWalk for home and community use, so that exoskeletons can be improved in the future to maximize their benefit to people with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* non-progressive spinal cord injury ≥1 year post-injury
* Body height between 5'3" and 6'4"
* Body weight ≤82 kg
* Uses wheelchair as primary mode of mobility
* If able to walk, walks at ≤0.4 m/s
* Arm strength sufficient to control forearm crutches
* Agree to attend intensive training of 1.5 hr/day, 4 days/wk for 14 weeks, plus testing pre and post training of approximately 2 weeks each

Exclusion Criteria:

* Contractures at the hip, knee or ankle that interferes with fitting into the ReWalk
* Fractures within the last 2 years
* Osteoporosis in the legs (t-score ≤-3.0)
* Severe postural hypotension
* Severe spasticity that interferes with use of the ReWalk
* Active pressure sores
* Pregnancy
* Severe head injury
* Conditions that preclude intensive exercise (such as high blood pressure)
* Presence of conditions contraindicated for transcranial magnetic stimulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2018-08-20 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaynie F Yang, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan AS, Livingstone DC, Hurd CL, Duchcherer J, Misiaszek JE, Gorassini MA, Manns PJ, Yang JF. Retraining walking over ground in a powered exoskeleton after spinal cord injury: a prospective cohort study to examine functional gains and neuroplasticity. J Neuroeng Rehabil. 2019 Nov 21;16(1):145. doi: 10.1186/s12984-019-0585-x. PMID 31752911
- [Derived] Manns PJ, Hurd C, Yang JF. Perspectives of people with spinal cord injury learning to walk using a powered exoskeleton. J Neuroeng Rehabil. 2019 Jul 19;16(1):94. doi: 10.1186/s12984-019-0565-1. PMID 31324256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 2014 to September 26, 2018. Recruitment was through previous contacts, word of mouth and SCI Alberta newsletter.
Period: Overall Study
Arm/Group | ReWalk Training
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All participants who completed mid point tests.
Arm/Group | ReWalk Training
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 11

OUTCOME MEASURES:

1. Primary Outcome: Physiological Cost Index (PCI) Ratio
Description: PCI is defined as the change in heart rate from the average at rest to the average in the last two minutes of the 6 minute walk test is divided by the average speed during the last two minutes of walking to give a measure of heartbeats/minute.
  The ratio between this measure while walking in the Rewalk and the same measure while performing the test using a wheelchair will be calculated. (Walk/wheelchair)
Time Frame: End of training:12-14 weeks from baseline
Population: Participants who completed 12 weeks of training intervention
Measure: Mean (Standard Deviation); unit: unit less
Arm/Group | ReWalk Training
Number analyzed (Participants) | 10
unit less | 3.34 (1.75)

2. Secondary Outcome: 10 Meter Walk Test
Description: Walking is timed over a 10 m section while the participant walks in the ReWalk in a 40 m hallway at the fastest safe speed possible.
Time Frame: End of training (at 12 weeks for 10 participants and 6 weeks for 1) and at follow-up (2-3 months from end of training)
Population: All participants who completed >6 weeks of training
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | ReWalk Training
Number analyzed (Participants) | 11
meters/second
  End of training | 0.41 (0.12)
  Follow-up: number analyzed (Participants) | 8
  Follow-up | 0.42 (0.10)

3. Secondary Outcome: Max Distance
Description: The maximum distance walked without a rest for up to one hour.
Time Frame: End of training:12-14 weeks from baseline
Population: Participants who completed 12 weeks of training
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | ReWalk Training
Number analyzed (Participants) | 10
meters | 1309 (457)

4. Secondary Outcome: Limits of Stability - Sitting
Description: While sitting/standing on a force plate, the participant will lean in 8 directions guided by a computer screen with feedback of the center of pressure. The sum of the maximum fore-aft and left right excursions was calculated. The changes from baseline to mid point of training, the end of the training phase (12 weeks) were calculated.
Time Frame: Baseline, Mid point-6 weeks from baseline, End training:12-14 weeks from baseline
Population: Participants able to sit unsupported at baseline and 12 weeks of training
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ReWalk Training
Number analyzed (Participants) | 10
cm
  Change at midpoint | 1.6 (2.6)
  Change at end of training | 4.5 (4.1)

5. Secondary Outcome: Sitting Sway
Description: Participants will sit on a force plate with feet unsupported, arms crossed over the chest and eyes closed. The trajectory of the center of pressure is measured for a maximum of 30 seconds or until balance is lost.
Time Frame: Baseline, Mid-point:6 weeks from baseline, End training:12-14 weeks from baseline
Population: Participants able to sit unsupported for greater than 22 seconds at baseline and after 12 weeks of training
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | ReWalk Training
Number analyzed (Participants) | 8
cm/s
  Change at midpoint | -1.59 (1.85)
  Change at end training | -1.38 (1.38)

6. Secondary Outcome: McGill Pain Questionnaire
Description: Paper/pencil questionnaire in which participant selects words that describe current pain. Words are divide into 20 subgroups and ranked within each group. A total score is tabulated by adding the number associated with the highest ranking word from each subgroup. Score range is from 0 to 73 with higher scores indicating greater pain.
Time Frame: Baseline, midpoint:6 weeks from baseline, end training:12-14 weeks from baseline
Population: Participants with neuropathic pain at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ReWalk Training
Number analyzed (Participants) | 9
score on a scale
  Baseline | 14.4 (11.4)
  Midpoint | 16.2 (11.7)
  End training | 11.1 (5.6)

7. Secondary Outcome: Spinal Cord Assessment Tool for Spastic Reflexes (SCATS)
Description: Response to 3 standardized tests: stretch of ankle plantarflexors, pin prick to the sole of the foot, stretch of the hip and knee flexors scored from 1 to 3. The scores form both lower extremities were summed (total score: no spasticity = 0; maximum spasticity = 36
Time Frame: Baseline, midpoint:6 weeks from baseline, end training:12-14 weeks from baseline
Population: Participants measured weekly for 12 weeks. P1 and P2 were measured only at baseline, 6 weeks and 12 weeks of training. P5 withdrew after 6 weeks of training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ReWalk Training
Number analyzed (Participants) | 8
score on a scale
  Baseline | 5.91 (6.17)
  Midpoint | 5.57 (4.35)
  End training | 6.25 (7.11)

8. Secondary Outcome: Motor Evoked Potentials
Description: Single pulse transcranial magnetic stimulation is delivered over the vertex to induce motor evoked potentials in the back extensor muscles. Electrical responses in paraspinal muscles were recorded at 8 levels spanning the injury. The peak to peak amplitude of the response was averaged over rials with background muscle contraction of 10 to 40 microvolts
Time Frame: Baseline, End training:12-14 weeks from baseline
Population: Participants with adequate background emg
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | ReWalk Training
Number analyzed (Participants) | 7
microvolts
  Baseline | 402 (193)
  End training | 353 (118)

9. Secondary Outcome: Change From Baseline in Manual Muscle Test at End of Training
Description: Five muscle groups in each lower extremity (hip flexors, knee extensors, ankle dorsiflexors, extensor of the big toe, and ankle plantarflexors) were tested as per the American Spinal Injury Association Impairment scale. Each muscle group was scored on a scale ranging from 0-5, where 0/5 indicates no muscle activity and is the lowest score and is considered to be a worse outcome. A score of 5/5 indicates normal strength and is considered the better outcome. The scores for all 10 muscle groups were summed so that the maximum score is 50. Change from baseline in Manual Muscle Test to end of training was calculated.
  0= total paralysis
  1. palpable or visible contraction
  2. active movement, gravity eliminated
  3. active movement, against gravity
  4. active movement, against some resistance
  5. active movement, against full resistance
Time Frame: Baseline, end training:12 -14 weeks from baseline
Population: Participants who completed 12 weeks of training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ReWalk Training
Number analyzed (Participants) | 10
units on a scale | 0.4 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of training (12 to 14 weeks from baseline).
Arm/Group | ReWalk Training
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReWalk Training (N=12)
Skin abrasion (Skin and subcutaneous tissue disorders) | 5 (12) — Abrasion to skin due to friction from device

LIMITATIONS AND CAVEATS:
Small number of participants suggests data should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT02322125/Prot_SAP_000.pdf